CLINICAL TRIAL: NCT05613907
Title: Can a Dedicated Chronic Limb-threatening Ischaemia (CLTI) Clinic Improve Patient Self
Brief Title: Can a Dedicated Chronic Limb-threatening Ischaemia (CLTI) Clinic Improve Patient Self-reported Quality of Life
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: VS22/151953
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Chronic Limb Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLTI clinic patients: This is a repeated measures study design. Eligible patients are opportunistically recruited into the study, and if successfully enrolled are given the EuroQoL 5-D to complete.
  Whether they undergo a revascularization procedure or not, the EuroQol 5-D is administered again at 6-12 weeks and again at 1 year after their initial assessment
  Interventions: Other: CLTI Clinic

INTERVENTIONS:
Other: CLTI Clinic — This is a specialist clinic designed to assess and manage patients with CLTI. Patients are assessed and imaged, and undergo elective revascularization procedures if appropriate

SUMMARY:
CLTI is the most severe form of peripheral arterial disease. Patients with the condition require investigation and management (typically in the form of revascularisation surgery) to salvage the limb. Traditionally, patients with the condition are admitted into hospital for their management, but with the advent of regional vascular networks, this is becoming increasingly difficult.

Recently, the Vascular Society of Great Britain and Ireland have advocated for the use of dedicated CLTI clinics to overcome this problem. Whilst there is burgeoning evidence for their clinical benefit, there is a lack of patient reported outcomes to measure their impact on patient selr-reported quality of life. We would like to determine if this service benefits its users as much as the clinical outcomes suggest it does.

DETAILED DESCRIPTION:
Chronic limb-threatening ischaemia (CLTI) is the most severe form of peripheral arterial disease (PAD). It affects 1% of the population and its incidence is expected to rise. It is a condition where the circulation to one, or both limbs is inadequate. It requires investigation and may require surgery in order to improve the blood flow to the affected limb(s). Without improvement in circulation, ulcers and gangrene set in, and the only cure is a major limb amputation.

Vascular surgery units in the United Kingdom have undergone centralisation into regional networks over the last decade in order to consolidate vascular surgery into 'high volume centres' to provide high quality care and better outcomes for patients.

However, national analysis of the performance of units has demonstrated that only 50% of CLTI patients are revascularised within the 'deliberately-challenging timeline' issued by the Vascular Society of Great Britain and Ireland (Birmpili et al., 2021; Vascular Society of Great Britain and Ireland, 2019).

CLTI already comprises more than 50% of vascular unit workload and the prevalence of CLTI is expected to rise, further increasing the burden on vascular services (Fowkes et al., 2016; Vascular Society of Great Britain and Ireland, 2018, 2021).

There is ample evidence demonstrating a strong inverse correlation between the provision of specialist outpatient clinics in the assessment and management of diabetic foot ulcers and major lower limb amputation (Joret et al., 2019; M Kerr, Rayman, & Jeffcoate, 2014; Marion Kerr, 2017; Monteiro-soares, Vale-lima, Martiniano, Dias, & Boyko, 2021; Paisey et al., 2017), Diabetic foot ulceration is a condition which has significant overlap with CLTI. It could therefore be inferred that a similar service for CLTI patients would also confer the same benefits.

At the Leeds Vascular Institute, we have implemented a dedicated CLTI clinic to assess and manage patients with the condition. Whilst there is limited evidence that these rapid access clinics can facilitate review and management of the condition, thereby successfully preventing major amputation in CLTI patients, the results are typically from single centre data series (Khan et al., 2020; Nickinson et al., 2021).

There is a paucity of evidence evaluating patient experience of this type of service. Therefore, the purpose of this study is to collect patient-reported outcome measure data at serial points in time, to determine whether a dedicated CLTI clinic can provide a significant and sustained improvement in self-reported quality of life for patients who utilise the service.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen and assessed in the CLTI clinic

Exclusion Criteria:

* Patients without a confirmed diagnosis of CLTI
* Patients with chronic venous insufficiency
* Patients with diabetic foot infection
* Patients with significant cognitive impairment such that they are unable to answer the questions

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up of opportunistic patients obtained from the CLTI clinic attendance register. They have been referred to the service either because they have a confirmed diagnosis of CLTI and need further management or the disease is suspected. Patients who do not have CLTI will be excluded as will those who do not have the ability to answer questions about their perceived quality of life
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assad Khan, BMBS, Principal Investigator — Leeds Vascular Institute, Leeds General Infirmary, Great George Street, Leeds, West Yorkshire, LS1 3EX, UK
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro-Soares M, Vale-Lima J, Martiniano J, Pinheiro-Torres S, Dias V, Boyko EJ. A systematic review with meta-analysis of the impact of access and quality of diabetic foot care delivery in preventing lower extremity amputation. J Diabetes Complications. 2021 Apr;35(4):107837. doi: 10.1016/j.jdiacomp.2020.107837. Epub 2020 Dec 31. PMID 33423910
- [Background] Paisey RB, Abbott A, Levenson R, Harrington A, Browne D, Moore J, Bamford M, Roe M; South-West Cardiovascular Strategic Clinical Network peer diabetic foot service review team. Diabetes-related major lower limb amputation incidence is strongly related to diabetic foot service provision and improves with enhancement of services: peer review of the South-West of England. Diabet Med. 2018 Jan;35(1):53-62. doi: 10.1111/dme.13512. Epub 2017 Oct 11. PMID 29023974
- [Result] Li Q, Birmpili P, Johal AS, Waton S, Pherwani AD, Boyle JR, Cromwell DA. Delays to revascularization for patients with chronic limb-threatening ischaemia. Br J Surg. 2022 Jul 15;109(8):717-726. doi: 10.1093/bjs/znac109. PMID 35543274
- [Result] Khan A, Hughes M, Ting M, Riding G, Simpson J, Egun A, Banihani M. A 'hot clinic' for cold limbs: the benefit of urgent clinics for patients with critical limb ischaemia. Ann R Coll Surg Engl. 2020 Jul;102(6):412-417. doi: 10.1308/rcsann.2020.0068. Epub 2020 Apr 20. PMID 32306742
- [Result] Nickinson ATO, Dimitrova J, Houghton JSM, Rate L, Dubkova S, Lines H, Gray LJ, Nduwayo S, Payne TJ, Sayers RD, Davies RSM. Does the Introduction of a Vascular Limb Salvage Service Improve One Year Amputation Outcomes for Patients with Chronic Limb-Threatening Ischaemia? Eur J Vasc Endovasc Surg. 2021 Apr;61(4):612-619. doi: 10.1016/j.ejvs.2020.12.007. Epub 2021 Feb 12. PMID 33583708

RESULTS

PARTICIPANT FLOW:
Groups:
- CLTI Clinic: This group comprises patients who have been referred into the CLTI clinic service prior to their first assessment. These patients will be given a structured outcome questionnaire like the EuroQoL 5D questionnaire that asks them to describe their symptoms.
  Whether they have revascularisation surgery or not, they are provided with a further EuroQoL 5-D questionnaire at 6-12 weeks and a final EuroQoL 5-D questionnaire at 1 year after their initial CLTI appointment
  CLTI Clinic: This is a specialist clinic designed to assess and manage patients with CLTI.
Period: Overall Study
Arm/Group | CLTI Clinic
Started | 30
Completed | 20
Not Completed | 10
Not completed — Lost to Follow-up | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- CLTI Clinic Patients: This is a repeated measures study design. Eligible patients are opportunistically recruited into the study, and if successfully enrolled are given the EuroQoL 5-D to complete.
  Whether they undergo a revascularization procedure or not, the EuroQol 5-D is administered again at 6-12 weeks and again at 1 year after their initial assessment
  CLTI Clinic: This is a specialist clinic designed to assess and manage patients with CLTI. Patients are assessed and imaged, and undergo elective revascularization procedures if appropriate
Arm/Group | CLTI Clinic Patients
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: EuroQoL-5D Visual Acuity Scale (VAS) Score
Description: The EuroQoL-5D is comprised of 2 parts, and the primary outcome involve scrutiny of the Visual Acuity Scale (VAS) represents a scale from 0 to 100 on which patients can report their own quality of life (0 the worst, 100 the best). The score is an integer and is measured again at 6-12 weeks, and again at 1-year post-initial assessment
Time Frame: Baseline - 6-12 weeks - 1-year
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CLTI Clinic Patients at Baseline: This is a repeated measures study design. Eligible patients are opportunistically recruited into the study, and if successfully enrolled are given the EuroQoL 5-D to complete, whether they undergo revascularisation or not.
  These are the results obtained at baseline
  CLTI Clinic: This is a specialist clinic designed to assess and manage patients with CLTI. Patients are assessed and imaged, and undergo elective revascularization procedures if appropriate
- CLTI Patients at 6-12 Weeks; CLTI Patients at 1-year: This is a repeated measures study design. Eligible patients are opportunistically recruited into the study, and if successfully enrolled are given the EuroQoL 5-D to complete, whether they undergo revascularisation or not.
  These are the results obtained between 6-12 weeks
  CLTI Clinic: This is a specialist clinic designed to assess and manage patients with CLTI. Patients are assessed and imaged, and undergo elective revascularization procedures if appropriate
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 6-12 Weeks | CLTI Patients at 1-year
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 47.55 (25.45) | 69.15 (14.16) | 65.35 (15.86)
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 6-12 Weeks; Test type: Superiority; p = 0.005, ANOVA; Mean Difference (Net) = -21.60, 95% CI 2-sided [-37.050 to -6.150], Standard Error of Mean 5.885
Statistical Analysis 2: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1-year; Test type: Superiority; p = 0.040, ANOVA; Mean Difference (Net) = -17.80, 95% CI 2-sided [-34.895 to -0.705], Standard Error of Mean 6.512
Statistical Analysis 3: Comparison: CLTI Patients at 6-12 Weeks vs CLTI Patients at 1-year; Test type: Superiority; p = 0.940, ANOVA; Mean Difference (Net) = 3.800, 95% CI 2-sided [-5.829 to 13.429], Standard Error of Mean 3.668

2. Secondary Outcome: EuroQoL-5D Movement
Description: The EuroQol-5D is comprised of 2 parts, and the secondary outcomes involve scrutiny of the separate QoL domains that give rise to the 5D in the name, which are: mobility; self-care; usual activities; pain; anxiety and depression. Patients self-report their own experiences on a 5-point scale. We are comparing pre- and post-intervention levels of the above.
Time Frame: At baseline and 1-year
Measure: Count of Participants; unit: Participants
Groups:
- CLTI Patients at 1 Year: This is a repeated measures study design. Eligible patients are opportunistically recruited into the study, and if successfully enrolled are given the EuroQoL 5-D to complete, whether they undergo revascularisation or not.
  These are the results obtained at 1 year
  CLTI Clinic: This is a specialist clinic designed to assess and manage patients with CLTI. Patients are assessed and imaged, and undergo elective revascularization procedures if appropriate
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 1 Year
Number analyzed (Participants) | 20 | 20
Participants
  No problems with mobility | 0 | 2
  Slight problems with mobility | 2 | 4
  Moderate problems with mobility | 7 | 6
  Severe problems with mobility | 11 | 7
  Unable to mobilise | 0 | 1
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1 Year; The null hypothesis is that there will be no significant difference in the EuroQol 5-D domains at 1 year compared to baseline; Test type: Superiority; p = 0.388, Wilcoxon Signed Ranks; Z statistic = -0.862

3. Secondary Outcome: EuroQoL-5D Self Care
Description: as for outcome 2
Time Frame: Baseline and 1-year
Measure: Count of Participants; unit: Participants
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 1 Year
Number analyzed (Participants) | 20 | 20
Participants
  No problems with self-care | 8 | 9
  Slight problems with self-care | 4 | 4
  Moderate problems with self-care | 4 | 4
  Severe problems with self-care | 4 | 2
  Unable to care for self | 0 | 1
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1 Year; The null hypothesis is that there will be no statistical difference in patient self-reported ability to perform basic self-care; Test type: Superiority; p = 0.974, Wilcoxon signed rank; Z statistic = -0.033

4. Secondary Outcome: EuroQoL 5-D Usual Activities
Description: as for outcome 2
Time Frame: Baseline and 1-year
Measure: Count of Participants; unit: Participants
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 1 Year
Number analyzed (Participants) | 20 | 20
Participants
  No problems performing usual activities | 2 | 6
  Slight problems performing usual activities | 4 | 5
  Moderate problems with performing usual activities | 6 | 7
  Severe problems with performing usual activities | 6 | 0
  I am unable to perform my usual activities | 2 | 2
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1 Year; The null hypothesis is no improvement in ability to perform usual activities at 1 year; Test type: Superiority; p = 0.118, Wilcoxon signed rank; Z statistic = -1.564

5. Secondary Outcome: EuroQoL 5-D Pain
Description: as for outcome 2
Time Frame: Baseline and 1-year
Measure: Count of Participants; unit: Participants
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 1 Year
Number analyzed (Participants) | 20 | 20
Participants
  No pain | 1 | 9
  Mild pain | 2 | 4
  Moderate pain | 6 | 3
  Severe pain | 10 | 3
  Extreme pain | 1 | 1
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1 Year; Test type: Superiority; p = 0.018, Wilcoxon signed rank; Z statistic = -2.364

6. Secondary Outcome: EuroQoL 5-D Anxiety and/or Depression
Description: as for outcome 2
Time Frame: Baseline and 1-year
Measure: Count of Participants; unit: Participants
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 1 Year
Number analyzed (Participants) | 20 | 20
Participants
  No anxiety and/or depression | 5 | 10
  Slight anxiety and/or depression | 6 | 1
  Moderate anxiety and/or depression | 6 | 9
  Severe anxiety and/or depression | 3 | 0
  Extreme anxiety and/or depression | 0 | 0
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1 Year; Test type: Superiority; p = 0.190, Wilcoxon signed rank — The null hypothesis is that there will be no difference in anxiety and/or depression compared to the initial visit; Z statistic = -1.311

7. Post Hoc Outcome: Revascularised EuroQoL 5-D VAS Score
Description: The EuroQoL-5D is comprised of 2 parts, and the primary outcome involve scrutiny of the Visual Acuity Scale (VAS) represents a scale from 0 to 100 on which patients can report their own quality of life (0 the worst, 100 the best). The score is an integer and is measured again at 6-12 weeks, and again at 1-year post-initial assessment.
  This sub-group analysis is of patients who underwent revascularisation procedures.
Time Frame: Baseline - 6-12 weeks - 1-year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 6-12 Weeks | CLTI Patients at 1-year
Number analyzed (Participants) | 13 | 13 | 13
score on a scale | 39.85 (27.525) | 66.69 (15.206) | 67.46 (16.008)
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 6-12 Weeks; Test type: Superiority; p = 0.027, ANOVA; Mean Difference (Net) = -26.846, 95% CI 2-sided [-50.762 to -2.390], Standard Error of Mean 8.604
Statistical Analysis 2: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1-year; Test type: Superiority; p = 0.024, ANOVA; Mean Difference (Net) = -27.615, 95% CI 2-sided [-51.837 to -3.394], Standard Error of Mean 8.715
Statistical Analysis 3: Comparison: CLTI Patients at 6-12 Weeks vs CLTI Patients at 1-year; Test type: Superiority; p = 1.000, ANOVA; Mean Difference (Net) = -0.769, 95% CI 2-sided [-13.374 to 11.836], Standard Error of Mean 4.535

8. Post Hoc Outcome: Non-operative EuroQoL 5-D VAS Score
Description: The EuroQoL-5D is comprised of 2 parts, and the primary outcome involve scrutiny of the Visual Acuity Scale (VAS) represents a scale from 0 to 100 on which patients can report their own quality of life (0 the worst, 100 the best). The score is an integer and is measured again at 6-12 weeks, and again at 1-year post-initial assessment.
  This sub-group analysis is of patients who did not undergo revascularisation procedures.
Time Frame: Baseline - 6-12 weeks - 1-year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLTI Clinic Patients at Baseline | CLTI Patients at 6-12 Weeks | CLTI Patients at 1-year
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 58.83 (12.954) | 73.71 (11.615) | 61.43 (15.999)
Statistical Analysis 1: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 6-12 Weeks; Test type: Superiority; p = 0.048, ANOVA; Mean Difference (Net) = -14.27, 95% CI 2-sided [-37.050 to -6.150], Standard Error of Mean 4.052
Statistical Analysis 2: Comparison: CLTI Clinic Patients at Baseline vs CLTI Patients at 1-year; Test type: Superiority; p = 1.000, ANOVA; Median Difference (Final Values) = -3.12, 95% CI 2-sided [-12.893 to 13.751], Standard Error of Mean 3.751
Statistical Analysis 3: Comparison: CLTI Patients at 6-12 Weeks vs CLTI Patients at 1-year; Test type: Superiority; p = 0.163, ANOVA; Mean Difference (Net) = 12.26, 95% CI 2-sided [-4.762 to 29.333], Standard Error of Mean 5.186

ADVERSE EVENTS:
Time Frame: 1 year
Description: Because this is a qualitative study where patients are provided a questionnaire. There is no exposure to risk for patients filling in a questionnaire
Arm/Group | CLTI Clinic
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Low recruitment numbers. This is multifactorial.

* Some patients feel unable to meaningfully answer the questions or engage with technology used to complete the questionnaire
* Some have mild memory impairment, and may struggle answering questions or remembering that they are enrolled.
* Some patients report felt overwhelmed by the diagnosis and management and either declined to participate or withdrew midway.
* CLTI is a condition with high mortality, and some patients did not survive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05613907/Prot_000.pdf
  • Informed Consent Form (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05613907/ICF_001.pdf